CLINICAL TRIAL: NCT06669741
Title: Clinical Outcomes Related to Arthroscopic Rotator Cuff Repair Recovery Using Semiconductor Embedded Therapeutic Garments From Incrediwear
Brief Title: Clinical Outcomes Related to Arthroscopic Rotator Cuff Repair Recovery Using Incrediwear
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Bone and Joint (Other)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Principal Investigator, Christopher Flowers, MD, Orthopaedic Surgeon, Texas Bone and Joint
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRBNet 2246455-1
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Arthropathy of Left Shoulder (Disorder); Rotator Cuff Arthropathy of Right Shoulder (Disorder); Rotator Cuff Arthropathy of Bilateral Shoulders
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-Controlled Clinical Investigation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): To assess the benefits of using the Incrediwear (Shoulder Sleeve) products for patients recovering from Arthroscopic Rotator Cuff Repair surgery for postoperative pain, range of motion, and swelling. We will compare patients with Incrediwear products or placebo Incrediwear products throughout a 12-week period with follow-ups up to 1-year post-surgery. The study will be double blinded as to the active Incrediwear sleeve vs placebo.
  Interventions: Device: Placebo
- Incrediwear Product (Active Comparator): To assess the benefits of using the Incrediwear (Shoulder Sleeve) products for patients recovering from Arthroscopic Rotator Cuff Repair surgery for postoperative pain, range of motion, and swelling. We will compare patients with Incrediwear products or placebo Incrediwear products throughout a 12-week period with follow-ups up to 1-year post-surgery. The study will be double blinded as to the active Incrediwear sleeve vs placebo.
  Interventions: Device: Shoulder Sleeve

INTERVENTIONS:
Device: Placebo — One group will receive placebo therapy (identical shoulder brace and arm sleeve absent of semiconductor fabric)
  Arms: Placebo
Device: Shoulder Sleeve — One group will receive active therapy (active semiconductor embedded shoulder brace and arm sleeve)
  Arms: Incrediwear Product

SUMMARY:
To assess the benefits of using the Incrediwear products for patients recovering from Arthroscopic Rotator Cuff Repair surgery for postoperative pain, range of motion, and swelling.

DETAILED DESCRIPTION:
Study Screening/pre-operative appointment

* The surgeon confirms the participant meets the inclusion criteria and is scheduled for surgery in the next few weeks.
* The surgeon will discuss the study and possible risks/benefits of being in the research.
* The study team will measure the participant wrist, arm, and shoulder circumference.
* The participant will rate their shoulder pain on a 1-10 Visual Analog Scale (VAS); shoulder function with the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire; shoulder function with the American Shoulder and Elbow Surgeons Score (ASES) scale, and function limitations using the Western Ontario Rotator Cuff Index (WORC) questionnaire.
* The study team will measure the patient's shoulder's range of motion, stability, and strength.
* Radiographic assessments may be analyzed if already indicated for patient care and included in standard of care procedure.

  • Day of Surgery
* A study packet will be given to the participant by the study staff. The packet will include a study number assignment, the products assigned, and the patient study journal. The participant, surgeon, and clinical staff will not know which group the participant is in.
* After surgery, the surgeon and PI, Dr. Flowers, will place the shoulder brace and arm sleeve according to the random assignment in the study packet. An abduction sling will then be placed on top of the shoulder brace and arm sleeve by Dr. Flowers.
* Participant will be instructed to wear the shoulder brace and arm sleeve for at least 20 hours per day, including overnight, for 12 weeks post-surgery.
* Participant will be instructed on the length of time to wear the shoulder abduction sling by the surgeon.
* The clinical staff will take arm circumference measurements post-surgery.

  • Postoperative Recovery: Weeks 1-12
* Follow-up visits will be at 2 weeks, 6 weeks, and 12 weeks post-surgery. During follow-up visits:

  * The clinical staff will take arm swelling measurements.
  * Participant shoulder pain on a 1-10 Visual Analog Scale (VAS); shoulder function with the Disabilities of the Arm, Shoulder, and Hand (DASH), American Shoulder and Elbow Surgeons score (ASES), and Western Ontario Rotator Cuff Index (WORC) questionnaires.
  * The clinical staff will measure shoulder's range of motion, stability, and strength.
  * Radiographic assessments may be analyzed if already indicated for patient care and included in standard of care procedure.
* Daily reported measures include:

  * Participant will record pain medication type and quantity taken in a medications log. Only medications related to the treatment of shoulder pain or function will be required to be reported.
  * Participant will rate shoulder pain severity on a 1-10 VAS in a pain diary log.
  * Participant will record how long they have worn the shoulder brace and arm sleeve in device usage log.
* At the 12th week follow-up visit all study products, including the shoulder brace, arm sleeve, medications log, pain diary log, and device usage log.

  • Postoperative Recovery: 6 months and 1 year post surgery
* A follow-up phone call after 6 months and 1-year post-surgery will be administered.
* Participant will be asked to rate shoulder pain on a 1-10 Visual Analog Scale (VAS) and shoulder function with the Disabilities of the Arm, Shoulder, and Hand (DASH), American Shoulder and Elbow Surgeons score (ASES), and Western Ontario Rotator Cuff Index (WORC) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing arthroscopic rotator cuff repair
2. Patients aged 18-75
3. Patients who are willing and able to adhere to follow-up schedule and protocol guidelines.
4. Patients who are willing and able to sign corresponding research subject consent form.

Exclusion Criteria:

1. Patient has a history of neurological conditions, including multiple sclerosis or Parkinson's disease
2. Patient has severe medical condition, including recent myocardial infarction, unstable angina, heart failure, severe anemia
3. Patient has had prior surgical treatment of a shoulder injury in the past 5 years
4. Patient has chronic pain conditions unrelated to shoulder condition
5. Patient has auto-immune or auto-inflammatory diseases
6. Patient has used tobacco within the last 90 days
7. Patient is not within the ages of 18-75
8. Patient has poorly controlled diabetes with HgA1c > 7.5
9. Patient has an active infection (local or systemic)
10. Patient is unwilling or unable to sign the corresponding research subject consent form
11. Patient meets any other criteria or has any other condition that, in the opinion of the investigator, would prevent them from completing the study or that, in the opinion of the investigator, would confound study results.
12. Against medical advice (AMA)
13. Prisoner as indicated in the medical record

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Arm Circumference Measure with a Measuring tape | Preop appointment, Postop Day 42, Day 84, Day 168, Day 364
  To measure swelling in the upper arm, a soft tape measure to measure the circumference of the arm at multiple points at the writs, mid-forearm, axilla, and oblique. A 2cm difference between arms at each area of the wrist, mid-forearm, axilla, and oblique shoulder is not optimal. Less than 2cm difference between arms at each area of the wrist, mid-forearm, axilla, and oblique shoulder is optimal.

SECONDARY OUTCOMES:
Visual Analogue Scale Measured by Scale | Preop appointment, Postop Day 42, Day 84, Day 168, Day 364
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The minimum number is zero meaning no pain and maximum number is 10 meaning the most pain the patient has every felt in their entire life. Lower scores are ideal while higher scores are indicative of the patient in a lot of pain.
Range of Motion Measured by a Goniometer | Preop appointment, Postop Day 42, Day 84, Day 168, Day 364
  To measure the range of motion of the shoulder, the patient will:
  Flexion: Move the arm forward and up until it's above the head. Extension: Move the arm backward. Abduction: Move the arm away from the body until it's above the head. Adduction: Move the arm toward the body. External rotation: With the elbow bent at a 90° angle, move the forearm away from the body.
  Internal rotation: With the elbow bent at a 90° angle, move the forearm toward the body.
  Shoulder flexion 0-180 degrees normal range Shoulder extension 0-60 degrees normal range Shoulder abduction 0-180 degrees normal range Shoulder adduction 180-0 degrees normal range Shoulder external rotation 0-90 degrees normal range Shoulder internal rotation 0-70 degrees normal range
  ...with lower number being poor and higher number being optimal

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L. Flowers, Principal Investigator — Texas Bone and Joint
Locations (1):
- Medical City Denton, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pre-approval to share data and data results must be obtained by the corporation.

REFERENCES:
- See also: Shoulder and Arm Sleeve — https://incrediwear.com/